CLINICAL TRIAL: NCT00022724
Title: Phase I/II Trial Of CCI-779 In Patients With Malignant Glioma
Brief Title: CCI-779 in Treating Patients With Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Purpose: Treatment
Other Study IDs: NABTC-0101; CDR0000068848 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Gliosarcoma | interventions — temsirolimus

INTERVENTIONS:
Drug: temsirolimus

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of CCI-779 in treating patients who have malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of CCI-779 in patients with malignant glioma.
* Determine the safety profile of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the efficacy of this drug, in terms of survival and objective response, in these patients.

OUTLINE: This is a dose-escalation study. Patients in phase II are stratified according to use of enzyme-inducing antiepileptic drugs (EIAEDs) (yes vs no) and disease type (glioblastoma multiforme with stable neuro-imaging after radiotherapy vs recurrent malignant glioma). Patients in phase I must be currently receiving EIAEDs.

* Phase I: Patients receive CCI-779 IV over 30 minutes once weekly. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of CCI-779 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive CCI-779 as in Phase I. Patients who are candidates for surgical resection of recurrent disease receive CCI-779 IV over 30 minutes 2 hours prior to surgery and then once weekly, as above, once recovered from surgery.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for phase I of this study within 12 months. A total of 87 patients will be accrued for phase II of this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed intracranial malignant glioma

  * Glioblastoma multiforme
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed oligoastrocytoma
  * Malignant astrocytoma not otherwise specified
* Initial diagnosis of low-grade allowed, if subsequently progressed
* Recurrent disease must have documented progression by MRI or CT scan
* Progressive disease must have failed prior radiotherapy
* Recent resection of recurrent or progressive tumor allowed provided all of the following are met:

  * Recovered from surgery
  * CT scan or MRI performed no more than 96 hours postoperatively OR at 4-6 weeks postoperatively
  * Concurrent steroid dosage must be stable
* Confirmation of true progressive disease (by PET, thallium scan, MR spectroscopy, or surgical documentation) required after prior interstitial brachytherapy or stereotactic radiosurgery

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 8 weeks

Hematopoietic:

* WBC at least 3,000/mm3
* Absolute neutrophil count at least 2,000/mm3
* Platelet count at least 120,000/mm3
* Hemoglobin at least 10 g/dL (transfusion allowed)

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT less than 1.5 times ULN
* Cholesterol less than 350 mg/dL
* Triglycerides less than 400 mg/dL

Renal:

* Creatinine less than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min

Other:

* No active infection
* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No significant medical illness that would preclude study
* No disease that would obscure toxicity or dangerously alter drug metabolism
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to CCI-779 or allergy to or inability to receive antihistamines
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 weeks after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior interferon

Chemotherapy:

* At least 2 weeks since prior vincristine
* At least 3 weeks since prior procarbazine
* At least 6 weeks since prior nitrosoureas
* Phase I:

  * 2 prior chemotherapy regimens allowed
  * 1 prior adjuvant regimen and 1 prior regimen for recurrent or progressive disease OR
  * 2 prior regimens for progressive tumor
* Phase II:

  * No more than 1 prior chemotherapy regimen for recurrent malignant glioma
  * No prior chemotherapy allowed for stable glioblastoma multiforme

Endocrine therapy:

* See Disease Characteristics
* At least 1 week since prior tamoxifen

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy for progressive disease
* No more than 1 month since prior radiotherapy for nonprogressive glioblastoma multiforme

Surgery:

* See Disease Characteristics

Other:

* Recovered from prior therapy
* At least 1 week since prior noncytotoxic agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2001-08-27 (Actual); Primary Completion 2006-05-04 (Actual); Study Completion 2007-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. Chang, MD, Study Chair — University of California, San Francisco
Locations (10):
- United States (10):
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Kuhn JG, Chang SM, Wen PY, Cloughesy TF, Greenberg H, Schiff D, Conrad C, Fink KL, Robins HI, Mehta M, DeAngelis L, Raizer J, Hess K, Lamborn KR, Dancey J, Prados MD; North American Brain Tumor Consortium and the National Cancer Institute. Pharmacokinetic and tumor distribution characteristics of temsirolimus in patients with recurrent malignant glioma. Clin Cancer Res. 2007 Dec 15;13(24):7401-6. doi: 10.1158/1078-0432.CCR-07-0781. PMID 18094423
- [Result] Chang SM, Wen P, Cloughesy T, Greenberg H, Schiff D, Conrad C, Fink K, Robins HI, De Angelis L, Raizer J, Hess K, Aldape K, Lamborn KR, Kuhn J, Dancey J, Prados MD; North American Brain Tumor Consortium and the National Cancer Institute. Phase II study of CCI-779 in patients with recurrent glioblastoma multiforme. Invest New Drugs. 2005 Aug;23(4):357-61. doi: 10.1007/s10637-005-1444-0. PMID 16012795
- [Result] Chang SM, Kuhn J, Wen P, Greenberg H, Schiff D, Conrad C, Fink K, Robins HI, Cloughesy T, De Angelis L, Razier J, Hess K, Dancey J, Prados MD; North American Brain Tumor Consortium And The National Cancer Institute. Phase I/pharmacokinetic study of CCI-779 in patients with recurrent malignant glioma on enzyme-inducing antiepileptic drugs. Invest New Drugs. 2004 Nov;22(4):427-35. doi: 10.1023/B:DRUG.0000036685.72140.03. PMID 15292713